CLINICAL TRIAL: NCT04538664
Title: A Randomized, Open-label Phase 3 Study of Combination Amivantamab and Carboplatin-Pemetrexed Therapy, Compared With Carboplatin-Pemetrexed, in Patients With EGFR Exon 20ins Mutated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Combination Amivantamab and Carboplatin-Pemetrexed Therapy, Compared With Carboplatin-Pemetrexed, in Participants With Advanced or Metastatic Non-Small Cell Lung Cancer Characterized by Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertions
Acronym: PAPILLON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108850; 61186372NSC3001 (Other: Janssen Research & Development, LLC); 2020-000633-40 (EudraCT Number); 2023-506033-29-00 (Registry Identifier: EUCT number)
Expanded Access: NCT04599712 (Approved for marketing)
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: EGFR Exon20ins Mutation; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Amivantamab + Chemotherapy (Experimental): Participants will receive pemetrexed 500 milligram per meter square (mg/m^2) intravenous (IV) infusion (with vitamin supplementation) on Day 1 of each 21-day cycle, in combination with carboplatin for up to 4 cycles, and then as maintenance monotherapy until disease progression. Carboplatin area under the concentration-time curve 5 milligram per milliliter (mg/mL) per minute (AUC 5) will be administered as IV infusion on Day 1 of each 21 day cycle, for up to 4 cycles. Participants will receive amivantamab 1400 mg (1750 mg if body weight is >=80 kilogram [kg]) by IV infusion once weekly up to Cycle 2 Day 1, then 1750 mg (2100 mg if body weight is >=80 kg) on Day 1 of each 21-day cycle, starting with Cycle 3. Following the primary analysis for efficacy, the study will transition to an OLE phase and participants will continue to receive the amivantamab plus chemotherapy in OLE phase. Participants who completed OLE period will enter LTE period and continue to receive same treatment.
  Interventions: Drug: Amivantamab; Drug: Pemetrexed; Drug: Carboplatin
- Arm B: Chemotherapy Alone (Experimental): Participants will receive pemetrexed 500 mg/m^2 IV infusion (with vitamin supplementation) on Day 1 of each 21-day cycle, in combination with carboplatin for up to 4 cycles, and then as maintenance monotherapy until disease progression. Carboplatin AUC 5 IV infusion will be administered on Day 1 of each 21-day cycle for up to 4 cycles. Following the primary analysis for efficacy, the study will transition to an OLE phase and participants will either continue to receive the chemotherapy or cross over to amivantamab in OLE phase. Participants who completed OLE period will enter LTE period and continue to receive same treatment.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be administered as an IV infusion at a dose of 1400 mg (1750 mg if body weight is >=80 kilogram [kg]) by once weekly up to Cycle 2 Day 1, then 1750 mg (2100 mg if body weight is >=80 kg) on Day 1 of each 21-day cycle, starting with Cycle 3 and will continue the same treatment in OLE phase then in LTE phase.
  Other Names: JNJ-61186372
  Arms: Arm A: Amivantamab + Chemotherapy
Drug: Pemetrexed — Pemetrexed will be administered as 500 mg/m^2 IV infusion (with vitamin supplementation) on Day 1 of each 21-day cycle and then as maintenance monotherapy until disease progression in Arm A and will continue the same treatment in OLE phase then in LTE phase.
  Arms: Arm A: Amivantamab + Chemotherapy
Drug: Carboplatin — Carboplatin will be administered as AUC 5 IV infusion for up to 4 cycles on Day 1 of each 21-day cycle.
Drug: Pemetrexed — Pemetrexed will be administered as 500 mg/m^2 IV infusion (with vitamin supplementation) on Day 1 of each 21-day cycle and then as maintenance monotherapy until disease progression in Arm B and will continue the same treatment in OLE phase then in LTE phase.
  Arms: Arm B: Chemotherapy Alone

SUMMARY:
The purpose of this study is to compare the efficacy, as demonstrated by progression-free survival (PFS), in participants treated with amivantamab in combination with chemotherapy, versus chemotherapy alone in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) characterized by EGFR Exon 20ins mutations.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically or cytologically confirmed, locally advanced or metastatic, nonsquamous non-small cell lung cancer (NSCLC) with documented primary epidermal growth factor receptor (EGFR) Exon 20ins activating mutation
* Participant must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Participant must agree to genetic characterization of tumor status through the required pretreatment tumor biopsy (or submission of equivalent archival material), as well as baseline and periodic blood samples for analysis of tumor mutations in the bloodstream
* A female participant of childbearing potential must have a negative serum or urine test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study

Exclusion Criteria:

* Participant has evidence of synchronous NSCLC disease (as suggested by genetic characterization or radiographic appearance)
* Participant has untreated brain metastases (a participant with definitively, locally treated metastases who is clinically stable, asymptomatic, and off corticosteroid treatment for at least 2 weeks prior to randomization is eligible)
* Participant has history of spinal cord compression that has not been treated definitively with surgery or radiation
* Participant has a medical history of interstitial lung disease (ILD), including drug-induced ILD, or radiation pneumonitis
* Participant has a contraindication to the use of carboplatin or pemetrexed (refer to local prescribing information for each agent). Participant has a history of hypersensitivity to, or cannot take, vitamin B12 or folic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2026-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (229):
- United States (17):
  - City of Hope, Duarte, California
  - University of California Irvine, Orange, California
  - UCLA, Santa Monica, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer & Research Institute, Tampa, Florida
  - University Cancer And Blood Center LLC, Athens, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University Medical Center, St Louis, Missouri
  - Regional Cancer Care Associates LLC, East Brunswick, New Jersey
  - Langone Health at NYC University, NYU School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Sanford Health, Sioux Falls, South Dakota
  - Texas Oncology Pa, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Blue Ridge Cancer Care, Salem, Virginia
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown
  - St George Hospital, Kogarah
  - Cabrini Medical Centre, Malvern
  - Sir Charles Gairdner Hospital, Nedlands
- Belgium (3):
  - UZ Leuven, Leuven
  - Algemeen Ziekenhuis Delta, Roeselare
  - CHU UCL Namur - Site Godinne, Yvoir
- Brazil (16):
  - Fundacao Pio XII, Barretos
  - Cetus Oncologia, Belo Horizonte
  - Ynova Pesquisa Clinica, Florianópolis
  - Oncosite - Centro de Pesquisa Clínica em Oncologia Ltda, Ijuí
  - Liga Norte Riograndense Contra O Cancer, Natal
  - UPCO Unidade de Pesquisa Clinica em Oncologia, Pelotas
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto D Or de Pesquisa e Ensino IDOR, Rio de Janeiro
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo
  - IOS - Instituto de Oncologia de Sorocaba Dr. Gilson Delgado, Sorocaba
  - Hospital Evangélico de Cachoeiro de Itapemirim, Vitória
- Canada (3):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- China (31):
  - Beijing Cancer Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Beijing Chest hospital, Capital medical university, Beijing
  - Peking University International Hospital, Beijing
  - Jilin cancer hospital, Changchun
  - Hunan Cancer hospital, Changsha
  - The First People's Hospital Of Changzhou, Changzhou
  - West China Hospital Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - The First Affiliated Hospital Zhejiang University College of Medicine, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Taizhou Hospital of Zhejiang Province, Linhai
  - Nanjing Drum Tower Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Cancer hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - Weifang People's Hospital, Weifang
  - TongJi Hospital of TongJi Medical College of Huazhong University of Science & Technology, Wuhan
  - Hospital of Jiangnan University, Wuxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
- France (9):
  - Institut Bergonie, Bordeaux
  - Hospices Civils de Lyon HCL, Bron
  - Centre Georges Francois Leclerc, Dijon
  - Centre Hospitalier Le Mans, Le Mans
  - CHR Hôpital Calmette, Lille
  - CHU Nantes - Hopital Nord Laënnec, Nantes
  - Institut Curie, Paris
  - CHU Bordeaux, Pessac
  - HIA Begin, Saint-Mandé
- Germany (10):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Kliniken der Stadt Koeln gGmbH, Cologne
  - Asklepios Klinik Gauting GmbH - Asklepios Fachkliniken Munchen-Gauting, Gauting
  - Thoraxklinik am Universitatsklinikum Heidelberg, Heidelberg
  - Onkologische Schwerpunktpraxis, Heilbronn
  - Bethanien Krankenhaus, Moers
  - Pius-Hospital Oldenburg, Oldenburg
  - Oncologianova GmbH, Recklinghausen
- Hungary (5):
  - Orszagos Koranyi Tbc es Pulmonologiai Intezet, Budapest
  - Mátrai Gyógyintézet-Bronchológia, Gyöngyös
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktatokorhaz, Székesfehérvár
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Tudogyogyintezet Torokbalint, Törökbálint
- India (6):
  - Basavatarakam Indo-American Hospital, Hyderabad
  - Tata Medical Center, Kolkata
  - Tata Memorial Hospital, Mumbai
  - HCG Manavta Cancer Centre, Nashik
  - Rajiv Gandhi Cancer Institute & Research Centre, New Delhi
  - Noble Hospital Pvt Ltd, Pune
- Israel (5):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - A O U Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliero Univ. Policlinico Gaspare Rodolico, Catania
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - San Gerardo Hospital, Monza
  - Ospedale S. Maria Delle Croci, Ravenna
  - Irccs Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (23):
  - Juntendo University Hospital, Bunkyō City
  - Saitama Medical University International Medical Center, Hidaka
  - National Hospital Organization Himeji Medical Center, Himeji
  - Kansai Medical University Hospital, Hirakata
  - Kanazawa University Hospital, Kanazawa
  - National Cancer Center Hospital East, Kashiwa
  - Kishiwada City Hospital, Kishiwada
  - Kobe City Medical Center General Hospital, Kobe
  - Kurashiki Central Hospital, Kurashiki
  - Kurume University Hospital, Kurume
  - Matsusaka Municipal Hospital, Matsusaka
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Kindai University Hospital, Osaka Sayama Shi
  - Kitasato University Hospital, Sagamihara
  - Hokkaido University Hospital, Sapporo
  - Iwate Medical University Hospital, Shiwa-gun
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Ehime University Hospital, Toon-shi
  - Wakayama Medical University Hospital, Wakayama
  - National Hospital Organization Yamaguchi Ube Medical Center, Yamaguchi
- Malaysia (4):
  - Hospital Pulau Pinang, George Town
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Mexico (8):
  - Centro Oncologico de Chihuahua, Chihuahua City
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Mexico Centre for Clinical Research, S.A. de C.V., Mexico City
  - Médica Sur, Mexico City
  - Instituto Nacional de Cancerologia, Mexico City
  - Health Pharma Professional Research, México
  - i Can Oncology Center, Monterrey
  - Oncologia Integral Satelite, Naucalpan
- Poland (6):
  - Centrum Onkologii im Prof F Lukaszczyka, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp z o o, Gdynia
  - Warminsko-Mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn
  - Private Specialist Hospitals - MedPolonia, Poznan
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Portugal (5):
  - Hosp. Cuf Descobertas, Lisbon
  - Uls Sao Jose - Hosp. Sto Antonio Dos Capuchos, Lisbon
  - Centro Hospitalar Universitario do Porto, EPE, Porto
  - Instituto Portugues de Oncologia, Porto
  - Centro Hospitalar de Vila Nova de Gaia Espinho E P E, Vila Nova de Gaia
- Pan American Center for Oncology Trials LLC, Rio Piedras, Puerto Rico
- Russia (13):
  - Irkutsk Regional Oncology Dispensary, Irkutsk
  - Moscow City Oncology Hospital № 62, Krasnogorsk
  - Krasnoyarsk Regional Oncology Dispensary, Krasnoyarsk
  - Leningrad Regional Oncology Dispensary, Kuzmolovsky
  - MCK, Moscow
  - City Clinical Hospital #1, Nal'chik
  - Nizhny Novgorod Regional Oncological Dispensary, Nizhny Novgorod
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Oncology Medical Clinics AV Medical group, Saint Petersburg
  - N.N. Petrov Research Institute Of Oncology, Saint Petersburg
  - Tomsk Cancer Research Institute, Tomsk
  - Bashkir State Medical University, Ufa
  - Yaroslavl Regional Clinical Oncology Hospital, Yaroslavl
- South Korea (11):
  - Inje University Haeundae Paik Hospital, Busan
  - National Cancer Center, Gyeonggi-do
  - GyeongSang National University Hospital, Gyeongsangnam-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (15):
  - Hosp Univ A Coruna, A Coruña
  - Inst. Cat. D'Oncologia-Badalona, Badalona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. Quiron Dexeus, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Burgos, Burgos
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp Virgen de La Victoria, Málaga
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
- Taiwan (6):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (3):
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Siriraj Hospital, Bangkok
  - Songklanagarind Hospital, Prince of Songkla University, Songkhla
- Turkey (Türkiye) (9):
  - Adana City Hospital, Adana
  - Başkent University Medical Faculty Adana Application and Research Center, Adana
  - Gazi University Hospital, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Trakya University Medical Faculty, Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Ic Hastaliklari Anabilim Dali Medikal Onkoloji Bd, Istanbul
  - Medipol Mega University Hospital, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Izmir Medical Park Hospital, Izmir
- Ukraine (3):
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk City Multifield Clinical Hospital # 4, Dnipro
  - Medical Center 'Ok Clinic' of LLC 'International Institute of Clinical Studies', Kyiv
  - National Cancer Institute, Kyiv
- United Kingdom (3):
  - Edinburgh Cancer Centre Western General, Edinburgh
  - The Royal Marsden NHS Trust, London
  - The Royal Marsden NHS Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Sanborn RE, Zhou C, Tang KJ, Cho BC, Cheng S, Popat S, Ono A, Lu S, Majem M, Aguilar A, Del Rosario Garcia Campelo M, Hayashi H, Lee KY, Lee SH, Delmonte A, Alatorre-Alexander J, Richardson G, Santos V, Dooms C, Sabari JK, Shu CA, Girard N, Mansfield AS, Park K, Xia Y, Bhattacharya A, Buyukkaramikli N, Perualila N, Diels J, Acharya S, Chandler C, Proskorovsky I, Dearden L, Wortman-Vayn H, Mahadevia PJ, Knoblauch RE, Agrawal T, Baig M, Felip E. Amivantamab-Chemotherapy in Non-Small Cell Lung Cancer with EGFR Exon 20 Insertions: Impact of Treatment Crossover and Other Endpoints from the Phase III PAPILLON Study. Target Oncol. 2025 Nov;20(6):979-989. doi: 10.1007/s11523-025-01182-0. Epub 2025 Nov 3. PMID 41184595
- [Derived] Kitazono S, Ono A, Kawamura T, Hataji O, Tanaka H, Matsumoto S, Watanabe N, Nagashima H, Oki M, Takahashi M, Anazawa T, Shirai T, Yamashita A, Wortman-Vayn H, Bhattacharya A, Agrawal T, Baig M, Knoblauch RE, Hayashi H. Amivantamab Plus Chemotherapy in Japanese Patients With EGFR Exon 20 Insertions NSCLC. Cancer Sci. 2025 Nov;116(11):3139-3148. doi: 10.1111/cas.70180. Epub 2025 Sep 8. PMID 40922529
- [Derived] Zhou C, Tang KJ, Cho BC, Liu B, Paz-Ares L, Cheng S, Kitazono S, Thiagarajan M, Goldman JW, Sabari JK, Sanborn RE, Mansfield AS, Hung JY, Boyer M, Popat S, Mourao Dias J, Felip E, Majem M, Gumus M, Kim SW, Ono A, Xie J, Bhattacharya A, Agrawal T, Shreeve SM, Knoblauch RE, Park K, Girard N; PAPILLON Investigators. Amivantamab plus Chemotherapy in NSCLC with EGFR Exon 20 Insertions. N Engl J Med. 2023 Nov 30;389(22):2039-2051. doi: 10.1056/NEJMoa2306441. Epub 2023 Oct 21. PMID 37870976

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Currently, the results are posted till cut-off date 03-May-2023. After completion of open-label extension (OLE) phase participant were allowed to enter the long-term extension (LTE) phase. LTE phase is still ongoing and results will be posted upon study completion.
Groups:
- Arm B: Chemotherapy Alone: Participants received chemotherapy with pemetrexed 500 milligrams per meter square (mg/m^2) Intraveous (IV) infusion (with vitamin supplementation) on Day 1 of each 21-day cycle, in combination with carboplatin area under the concentration-time curve of 5 (AUC 5) IV infusion administered on Day 1 for up to 4 cycles, and then as maintenance monotherapy until disease progression. Following the primary analysis, the study was transitioned to an open-label extension (OLE) phase, and participants either continued to receive the chemotherapy or crossover to amivantamab in the OLE phase.
- Arm A: Amivantamab + Chemotherapy: Participants received amivantamab 1400 milligrams (mg) (1750 mg if body weight is greater than or equal to (>=) 80 kilograms [kg]) by IV infusion once weekly starting from Cycle 1 Day 1 up to Cycle 2 Day 1, then 1750 mg (2100 mg if body weight is >=80 kg) on Day 1 of each 21-day cycle, starting with Cycle 3 up to Cycle 5 Day 1. Participants received chemotherapy with pemetrexed 500 mg/m^2 IV infusion (with vitamin supplementation) on Day 1 of each 21-day cycle, in combination with carboplatin area under the concentration-time curve of 5 milligrams per milliliter (mg/mL) per minute (AUC 5) was administered as an IV infusion on Day 1, for up to 4 cycles, and then as maintenance monotherapy until disease progression. Following the primary analysis, the study was transitioned to an OLE phase, and participants continued to receive amivantamab plus chemotherapy in the OLE phase.
Period: Overall Study
Arm/Group | Arm B: Chemotherapy Alone | Arm A: Amivantamab + Chemotherapy
Started | 155 | 153
Treated | 155 | 151
Completed (As per protocol, participants who died were also considered as completed.) | 42 | 28
Not Completed | 113 | 125
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Lost to Follow-up | 2 | 1
Not completed — Ongoing | 106 | 115

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm B: Chemotherapy Alone | Arm A: Amivantamab + Chemotherapy | Total
Number analyzed (Participants) | 155 | 153 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12.01) | 59.3 (11.92) | 59.6 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 85 | 178
  Male | 62 | 68 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 13 | 22
  Not Hispanic or Latino | 145 | 137 | 282
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 89 | 97 | 186
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 60 | 49 | 109
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 4 | 2 | 6
  BELGIUM | 1 | 2 | 3
  BRAZIL | 5 | 6 | 11
  CANADA | 3 | 5 | 8
  CHINA | 48 | 39 | 87
  FRANCE | 4 | 3 | 7
  GERMANY | 2 | 0 | 2
  HUNGARY | 0 | 1 | 1
  INDIA | 6 | 5 | 11
  ISRAEL | 2 | 1 | 3
  ITALY | 5 | 7 | 12
  JAPAN | 15 | 19 | 34
  MALAYSIA | 1 | 10 | 11
  MEXICO | 2 | 1 | 3
  POLAND | 2 | 4 | 6
  PORTUGAL | 3 | 1 | 4
  RUSSIAN FEDERATION | 3 | 0 | 3
  SOUTH KOREA | 10 | 13 | 23
  SPAIN | 13 | 16 | 29
  TAIWAN | 5 | 4 | 9
  THAILAND | 0 | 2 | 2
  TURKEY | 10 | 3 | 13
  UNITED KINGDOM | 3 | 1 | 4
  UNITED STATES | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization until the date of objective disease progression based on BICR using RECIST version 1.1 or death (by any cause) in the absence of progression, whichever came first. Participants who have not progressed or have not died at the time of analysis were censored at the time of the latest date of their last evaluable RECIST version 1.1 assessment. Pharmacodynamic: Sum of diameters increased by greater than or equal to (>=)20 percent (%) and >=5 millimeter (mm) from nadir (including baseline if it was smallest sum).
Time Frame: From randomization to either disease progression or death whichever occurs first (up to 29 months)
Population: Full analysis set included all randomized participants, classified according to their assigned treatment arm regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm B: Chemotherapy Alone | Arm A: Amivantamab + Chemotherapy
Number analyzed (Participants) | 155 | 153
Months | 6.70 [5.59 to 7.33] | 11.37 [9.79 to 13.70]
Statistical Analysis 1: Comparison: Arm B: Chemotherapy Alone vs Arm A: Amivantamab + Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.395, 95% CI 2-sided [0.296 to 0.528]

2. Secondary Outcome: Objective Response Rate (ORR)
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

3. Secondary Outcome: Duration of Response (DoR)
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

4. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

5. Secondary Outcome: Time to Subsequent Therapy (TST)
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

6. Secondary Outcome: Progression-Free Survival After First Subsequent Therapy (PFS2)
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

7. Secondary Outcome: Time to Symptomatic Progression (TTSP)
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

8. Secondary Outcome: Number of Participants Treatment-emergent Adverse Events (TEAEs)
Time Frame: From Day 1 to 5 years 2 months
Reporting Status: Not Posted, anticipated posting 2027-01

9. Secondary Outcome: Number of Participants TEAEs With Severity
Time Frame: From Day 1 to 5 years 2 months
Reporting Status: Not Posted, anticipated posting 2027-01

10. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

11. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

12. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Time Frame: Up to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

13. Secondary Outcome: Serum Concentration of Amivantamab
Time Frame: Day 1 (Cycles 1, 2, 3, 5, 7, 9, 11, 13), Day 2 (Cycle 1)
Reporting Status: Not Posted, anticipated posting 2027-01

14. Secondary Outcome: Number of Participants With Anti-Amivantamab Antibodies
Time Frame: Day 1 (Cycles 1, 2, 3, 5, 7, 9, 11, 13), Day 2 (Cycle 1)
Reporting Status: Not Posted, anticipated posting 2027-01

15. Secondary Outcome: Change From Baseline in European Organization of Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30)
Time Frame: From baseline to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

16. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurement Information System-Physical Function (PROMIS-PF)
Time Frame: From baseline to 5 years 3 months
Reporting Status: Not Posted, anticipated posting 2027-01

ADVERSE EVENTS:
Time Frame: From baseline (Day 1 of Cycle 1) up to 29 months
Description: The safety set included all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Arm B: Chemotherapy Alone | Arm A: Amivantamab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 42/155 | 28/151
Serious Adverse Events (participants affected / at risk) | 48/155 | 56/151
Other Adverse Events (participants affected / at risk) | 149/155 | 151/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm B: Chemotherapy Alone (N=155) | Arm A: Amivantamab + Chemotherapy (N=151)
Pneumonia (Infections and infestations) | 4 | 6
Covid-19 (Infections and infestations) | 1 | 3
Cellulitis (Infections and infestations) | 1 | 2
Rash Pustular (Infections and infestations) | 0 | 2
Skin Infection (Infections and infestations) | 0 | 2
Covid-19 Pneumonia (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Pneumonia Viral (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 6 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Myoclonic Epilepsy (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lacunar Infarction (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 0
Asthenia (General disorders) | 1 | 2
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 1
Blood Creatinine Increased (Investigations) | 1 | 1
C-Reactive Protein Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Endometrial Thickening (Reproductive system and breast disorders) | 0 | 1
Ovarian Mass (Reproductive system and breast disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Biliary Obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 1 | 0
Contrast Media Reaction (Immune system disorders) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm B: Chemotherapy Alone (N=155) | Arm A: Amivantamab + Chemotherapy (N=151)
Rash (Skin and subcutaneous tissue disorders) | 12 | 81
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 5 | 47
Dry Skin (Skin and subcutaneous tissue disorders) | 6 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 10
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 10
Erythema (Skin and subcutaneous tissue disorders) | 8 | 1
Constipation (Gastrointestinal disorders) | 47 | 60
Nausea (Gastrointestinal disorders) | 65 | 55
Stomatitis (Gastrointestinal disorders) | 9 | 38
Diarrhoea (Gastrointestinal disorders) | 19 | 31
Vomiting (Gastrointestinal disorders) | 28 | 31
Haemorrhoids (Gastrointestinal disorders) | 2 | 18
Mouth Ulceration (Gastrointestinal disorders) | 4 | 12
Abdominal Pain (Gastrointestinal disorders) | 4 | 10
Gingival Bleeding (Gastrointestinal disorders) | 2 | 8
Abdominal Distension (Gastrointestinal disorders) | 10 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 | 62
Decreased Appetite (Metabolism and nutrition disorders) | 43 | 54
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 32
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 | 22
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 19
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 10
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 8
Neutropenia (Blood and lymphatic system disorders) | 70 | 88
Anaemia (Blood and lymphatic system disorders) | 84 | 76
Leukopenia (Blood and lymphatic system disorders) | 50 | 56
Thrombocytopenia (Blood and lymphatic system disorders) | 46 | 55
Lymphopenia (Blood and lymphatic system disorders) | 11 | 7
Oedema Peripheral (General disorders) | 16 | 45
Asthenia (General disorders) | 28 | 29
Pyrexia (General disorders) | 9 | 24
Fatigue (General disorders) | 32 | 23
Malaise (General disorders) | 12 | 16
Mucosal Inflammation (General disorders) | 4 | 15
Oedema (General disorders) | 2 | 10
Paronychia (Infections and infestations) | 0 | 85
Covid-19 (Infections and infestations) | 20 | 33
Pneumonia (Infections and infestations) | 8 | 13
Conjunctivitis (Infections and infestations) | 7 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 9
Urinary Tract Infection (Infections and infestations) | 8 | 6
Alanine Aminotransferase Increased (Investigations) | 56 | 50
Aspartate Aminotransferase Increased (Investigations) | 50 | 47
Gamma-Glutamyltransferase Increased (Investigations) | 26 | 21
Weight Decreased (Investigations) | 13 | 21
Blood Alkaline Phosphatase Increased (Investigations) | 12 | 19
Blood Lactate Dehydrogenase Increased (Investigations) | 8 | 13
Blood Creatinine Increased (Investigations) | 14 | 11
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 | 63
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 16
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Dizziness (Nervous system disorders) | 15 | 15
Dysgeusia (Nervous system disorders) | 10 | 9
Headache (Nervous system disorders) | 13 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 16 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 10
Insomnia (Psychiatric disorders) | 20 | 16
Hyperbilirubinaemia (Hepatobiliary disorders) | 6 | 15
Deep Vein Thrombosis (Vascular disorders) | 3 | 10
Hypertension (Vascular disorders) | 10 | 1
Lacrimation Increased (Eye disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT04538664/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT04538664/SAP_001.pdf